CLINICAL TRIAL: NCT05254795
Title: Precision Medicine Randomized Clinical Trial Comparing Molecular Tumor Board Assisted Care to Usual Care
Acronym: PRiMAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Timothy Mullett (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Timothy Mullett, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MCC-21-LUN-126-PMC
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Molecular tumor board
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care recipients (No Intervention)
- Molecular tumor board intervention (Experimental)
  Interventions: Other: Molecular tumor board assisted care

INTERVENTIONS:
Other: Molecular tumor board assisted care — Participants in this group will obtain recommendations for care from the molecular tumor board.
  Arms: Molecular tumor board intervention

SUMMARY:
This trial will compare Molecular Tumor Board (MTB) assisted care to usual care for patients who have newly diagnosed histologically or cytologically confirmed stage IIb-IV Non-Small Cell Lung Cancer (NSCLC) and are planning to undergo treatment for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinically suspected or histologically confirmed stage IIb-IV NSCLC who are planning to undergo treatment
* No prior systemic therapies for NSCLC, with the exception of adjuvant therapy for early stage NSCLC. Prior surgery and/or radiation is allowed.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with targeted therapy, in the opinion of the treating physician.
* Pregnancy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Overall survival 1 year survival between individuals with stage IIb-IV NSCLC who receive MTB assisted care to those who receive usual care.
Change in quality of life (QOL) | At enrollment, 8 weeks, and 12 weeks.
  Quality of life will be assessed via the FACT-L (The Functional Assessment of Cancer Therapy - Lung). FACT-L has 5 areas of measurement: physical wellbeing, social/family wellbeing, emotional wellbeing, functional wellbeing, and an additional concerns list of problems specific to lung cancer. Areas are measured on a 5-point Likert-type scale of 0-4. The FACT-L subscales can be scored to yield a total score, subscale scores, as well as the Trial Outcome Index (TOI), which reflects the physical wellbeing, functional wellbeing, and lung cancer symptom subscales. TOI scores range from 0-84, with a higher score reflecting better QOL. Total FACT-G scores (physical, social, emotional, and functional wellbeing subscales) range from 0-108, with higher scores reflecting better QOL. The lung cancer subscale (i.e., additional concerns subscale) can range from 0-28 (only 7 items are scored), with higher scores reflecting better QOL.

SECONDARY OUTCOMES:
Overall survival | 1 year
  Comparison of overall survival between individuals with stage IIb-IV NSCLC who receive MTB assisted care to those who receive usual care
Change in guideline concordant care | 8 weeks, 12 weeks, and 1 year
  Comparison of guideline concordant care (specifically receiving next generation sequencing (NGS) testing and treatments based on identified mutations) between individuals with stage IIb-IV NSCLC who receive MTB assisted care to those who receive usual care.
Change in satisfaction with treatment | At enrollment, 8 weeks, and 12 weeks.
  To compare satisfaction with treatment between individuals with stage IIb-IV NSCLC who receive MTB assisted care to those who receive usual care, including financial, psychosocial, and physical measures of satisfaction using the Functional Assessment of Chronic Illness Therapy (FACIT) - Treatment Satisfaction - General (TSG) (version 4). The FACIT-TSG is an 8-item questionnaire, with each item score ranging from 0 ("not at all") to 4 ("very much"). Total scores range from 0 to 32 with higher scores indicating greater satisfaction with treatment.

OTHER OUTCOMES:
Association of ctDNA variant allele frequency | 1 year
  To determine the association of ctDNA variant allele frequency with 1 year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Mullett, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No